CLINICAL TRIAL: NCT01781468
Title: A Phase III Randomized, Double-Blind Placebo Controlled Study of Armodafinil (Nuvigil®) To Reduce Cancer-Related Fatigue in Patients With High Grade Glioma
Brief Title: Armodafinil in Reducing Cancer-Related Fatigue in Patients With High Grade Glioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A221101; N10C3; NCI-2012-02020 (Registry Identifier: Clinical Trial Reporting Program); U10CA037404 (NIH); U10CA037447 (NIH); UG1CA189823 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive 150 mg armodafinil orally every day in the morning for 8 weeks.
  Interventions: Drug: armodafinil 150 mg
- Arm II (Placebo Comparator): Patients receive placebo orally every day in the morning for 8 weeks.
  Interventions: Other: Placebo
- Arm III (Experimental): Patients receive 250 mg armodafinil orally every day in the morning for 8 weeks.
  Interventions: Drug: armodafinil 250 mg

INTERVENTIONS:
Drug: armodafinil 150 mg — given orally
  Arms: Arm I
Other: Placebo — given orally
  Arms: Arm II
Drug: armodafinil 250 mg — given orally
  Arms: Arm III

SUMMARY:
This randomized phase III trial studies armodafinil to see how well it works in reducing cancer-related fatigue in patients with high grade glioma. Armodafinil may help relieve fatigue in patients with high grade glioma.

DETAILED DESCRIPTION:
Patients experiencing fatigue related to cancer will be asked to take part in this study. Cancer-related fatigue is a very common symptom in patients with cancer. Patients will receive armodafinil or placebo. Please see the "Arms" section for more details regarding the treatment assignments. The primary objective of this study is to determine preliminary efficacy measured by patient reported fatigue Brief Fatigue Inventory (BFI) at 8 weeks of two doses (150 mg and 250 mg) of armodafinil in treating moderate fatigue compared to placebo in patients with high grade glioma.

The secondary objectives of the study are listed below.

1. To evaluate the tolerability at 8 weeks of 150 mg and 250 mg armodafinil in this patient population.
2. To assess the effect of armodafinil at 8 weeks on cognitive function in patients with high grade glioma.
3. To assess the impact of armodafinil on global quality of life and other fatigue endpoints in this patient population with high grade glioma.
4. Explore the correlation between the BFI, Patient-Reported Outcomes Measurement Information System (PROMIS), and Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) measures, as well as, the relationship of fatigue and cognitive difficulties.

Patients will receive armodafinil or placebo for a total of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with glioblastoma, gliosarcoma, small cell or large cell glioblastoma, glioblastoma with oligo features, glioblastoma with primitive neuroectodermal tumor-like components (GBM-PNET) features, anaplastic astrocytoma, anaplastic oligodendroglioma, or anaplastic oligoastrocytoma who are clinically stable and have completed radiation therapy (excluding stereotactic radiosurgery) > 21 days and =< 24 months prior to enrollment; NOTE: clinical stability will be defined as a stable or improved Karnofsky performance status (KPS) compared to the prior month
* >= 6 score on the worst fatigue question of the BFI (Brief Fatigue Inventory, question 3); it is not required for the patient to complete the entire BFI to meet this criterion
* Undergone surgery (gross total or subtotal resection) or biopsy and will have been treated with concurrent radiation therapy and chemotherapy as standard of care for glioblastoma, gliosarcoma, small cell or large cell glioblastoma, glioblastoma with oligo features, glioblastoma with primitive neuroectodermal tumor-like components (GBM-PNET) features, anaplastic astrocytoma, anaplastic oligodendroglioma, or anaplastic oligoastrocytoma patients; Note: radiation must be completed, but chemotherapy is allowed; patients who are currently using Optune device will be eligible to participate in this trial
* Negative serum pregnancy test done =< 7 days prior to registration only for women determined to be of childbearing potential by their treating physician
* Ability to complete questionnaire(s) by themselves or with assistance
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, 2 or 3
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Stable dose of corticosteroid >= 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2013-06-21 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyx B. Porter Umphrey, MD, Study Chair — Mayo Clinic
Locations (365):
- United States (365):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Memorial Medical Center, Modesto, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - The NeuroMedical Center-Clinic, Baton Rouge, Louisiana
  - Culicchia Neurological Clinic LLC, Marrero, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Unspecified Site, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - UP Health System Hematology Oncology Marquette, Marquette, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Freeman Health System, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University Radiation Oncology, Rochester, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint John Medical Center, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Thompson Oncology Group-Lenoir City, Lenoir City, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Austin Cancer Centers-Central Austin, Austin, Texas
  - Austin Cancer Centers-North, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in the publication PubMed ID 34882169.
Time Frame: The data underlying the publication is available as of 10/20/2023 and will be available for the duration of the NCTN/NCORP Data Archive. .
Access Criteria: Instructions
  1. Click to open the Protocol Section.
  2. Click Edit next to the IPD Sharing Statement and select options for "Plan to Share IPD".
  3. Click Edit next to the References section.
  4. Under the References section, edit the following fields:
     1. Links: https://nctn-data-archive.nci.nih.gov/
     2. Available IPD/Information: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Derived] Porter AB, Liu H, Kohli S, Cerhan JL, Sloan J, McMurray RP, Le-Rademacher J, Loprinzi CL, Villano JL, Kizilbash SH, Mehta MP, Jaeckle KA, Brown PD. Efficacy of Treatment With Armodafinil for Cancer-Related Fatigue in Patients With High-grade Glioma: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2022 Feb 1;8(2):259-267. doi: 10.1001/jamaoncol.2021.5948. PMID 34882169

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (150 mg Armodafinil): Patients receive 150 mg armodafinil orally every day in the morning for 8 weeks.
- Arm II (250 mg Armodafinil): Patients receive 250 mg armodafinil orally every day in the morning for 8 weeks.
- Arm III (Placebo): Patients receive placebo orally every day in the morning for 8 weeks.
Period: Overall Study
Arm/Group | Arm I (150 mg Armodafinil) | Arm II (250 mg Armodafinil) | Arm III (Placebo)
Started | 109 | 110 | 109
Completed (Evaluable for the Primary Endpoint) | 103 | 97 | 97
Not Completed | 6 | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (150 mg Armodafinil) | Arm II (250 mg Armodafinil) | Arm III (Placebo) | Total
Number analyzed (Participants) | 109 | 110 | 109 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.92) | 56.9 (12.21) | 56.6 (12.8) | 57.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 43 | 135
  Male | 63 | 64 | 66 | 193
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 101 | 105 | 104 | 310
  Race: Non-White | 8 | 5 | 5 | 18
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 18 | 28 | 23 | 69
    1 | 60 | 58 | 62 | 180
    2 | 23 | 22 | 16 | 61
    3 | 8 | 2 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Response in Terms of a Clinically Meaningful Improvement in Patient-reported Fatigue at 8 Weeks.
Description: A response is defined as an improvement of 2 points on the 0-10 scale of the usual fatigue on the Brief Fatigue Inventory (BFI). The number of participants with a response in terms of a clinically meaningful improvement in patient-reported fatigue at 8 weeks.
  Scale: 0 (No fatigue) - 10 (As bad as you can imagine) Interpretation: higher scores mean a worse outcome
Time Frame: At 8 weeks
Population: Participants who completed the study are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (150 mg Armodafinil) | Arm II (250 mg Armodafinil) | Arm III (Placebo)
Number analyzed (Participants) | 103 | 97 | 97
Participants | 29 | 27 | 29
Statistical Analysis 1: Comparison: Arm I (150 mg Armodafinil) vs Arm II (250 mg Armodafinil) vs Arm III (Placebo); Test type: Superiority; p = 0.9601, Fisher Exact

2. Secondary Outcome: Fatigue: Brief Fatigue Inventory (BFI): The Number of Participants With a Response in Terms of a Clinically Meaningful Improvement in Patient-reported Fatigue at 4 Weeks.
Description: A response is defined as an improvement of 2 points on the 0-10 scale of the usual fatigue on the Brief Fatigue Inventory (BFI). The number of participants with a response in terms of a clinically meaningful improvement in patient-reported fatigue at 4 weeks Scale: 0 (No fatigue) - 10 (As bad as you can imagine) Interpretation: higher scores mean a worse outcome
Time Frame: Up to 4 weeks
Population: Participants who completed the study are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (150 mg Armodafinil) | Arm II (250 mg Armodafinil) | Arm III (Placebo)
Number analyzed (Participants) | 103 | 97 | 97
Participants | 37 | 31 | 30
Statistical Analysis 1: Comparison: Arm I (150 mg Armodafinil) vs Arm II (250 mg Armodafinil) vs Arm III (Placebo); Test type: Superiority; p = 0.7877, Fisher Exact

3. Secondary Outcome: Cognitive Function: Assessed by the Change in Z Score for Symbol Digit Modalities Test (SDMT) From Baseline to End of Week 8
Description: The participant is presented with a page headed by a key that pairs the single digits 1-9 with nine symbols. Rows below contain only symbols, the subject's task is to orally report the correct number in the spaces below. After completing the first 10 items with guidance, the subject is timed to determine how many responses can be made in 90 seconds. Range score: not applicable. Higher scores mean a better outcome. Explored domain: Sustained attention and information processing speed. Each neuropsychological measure was converted to an age-normative z score using published normative data. Impaired SDMT performance was defined as falling one standard deviation or more below the normative mean.
Time Frame: Up to 8 weeks
Population: Participants who completed the Symbol Digit Modalities Test at baseline and end of week 8 are included in this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm I (150 mg Armodafinil) | Arm II (250 mg Armodafinil) | Arm III (Placebo)
Number analyzed (Participants) | 61 | 55 | 60
units on a scale | 0.0 [-1.6 to 2.5] | 0.3 [-3.4 to 2.5] | 0.0 [-3.4 to 4.9]
Statistical Analysis 1: Comparison: Arm I (150 mg Armodafinil) vs Arm II (250 mg Armodafinil) vs Arm III (Placebo); Test type: Superiority; p = 0.3272, Kruskal-Wallis

4. Secondary Outcome: Change in Quality of Life as Measured by Linear Analogue Self Assessment (LASA) From Baseline to End of Weeks 4 and 8
Description: Quality of life: Linear Analogue Self Assessment (LASA) will be analyzed comparing the total score for each treatment testing for change from baseline to four and eight weeks. Linear Analogue Self Assessment (LASA) is a 12 global QOL tool to which measures 10 subscales: overall QOL, physical well-being, fatigue, frequency and severity of pain, as well as social functioning and spiritual, emotional and mental well-being. All subscales were converted to a scale of 0-100, with higher scores indicating better QOL. Total score is the average of all 10 subscales.
Time Frame: Up to 8 weeks
Population: Participants with LASA data available at all specified time points are included in this analysis. The number analyzed in row differ from the Overall number of participants who completed the study due to missing data (i.e. participants did not complete the LASA at either week 4 and/or week 8 time point(s)).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm I (150 mg Armodafinil) | Arm II (250 mg Armodafinil) | Arm III (Placebo)
Number analyzed (Participants) | 80 | 68 | 84
units on a scale
  Baseline to Week 4 | 2.0 [-23.0 to 31.0] | 0.5 [-25.0 to 29.0] | 2.0 [-10.0 to 26.0]
  Baseline to Week 8: number analyzed (Participants) | 64 | 59 | 69
  Baseline to Week 8 | 4.0 [-32.0 to 26.0] | 3.0 [-16.0 to 27.0] | 2.0 [-15.0 to 27.0]
Statistical Analysis 1: Comparison: Arm I (150 mg Armodafinil) vs Arm II (250 mg Armodafinil) vs Arm III (Placebo); Baseline to Week 4; Test type: Superiority; p = 0.9122, Kruskal-Wallis
Statistical Analysis 2: Comparison: Arm I (150 mg Armodafinil) vs Arm II (250 mg Armodafinil) vs Arm III (Placebo); Baseline to Week 8; Test type: Superiority; p = 0.8559, Kruskal-Wallis

5. Secondary Outcome: Number of Participants Who Experienced at Least One Grade 3 or Higher Adverse Events Deemed at Least Possibly Related to Treatment Via the CTCAE Version 4.0
Description: The number of participants who experienced at least one grade 3 or higher adverse events deemed at least possibly related to treatment via the CTCAE version 4.0
Time Frame: Up to 8 weeks
Population: Participants who started the study are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (150 mg Armodafinil) | Arm II (250 mg Armodafinil) | Arm III (Placebo)
Number analyzed (Participants) | 109 | 110 | 109
Participants | 6 | 8 | 3

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | Arm I (150 mg Armodafinil) | Arm II (250 mg Armodafinil) | Arm III (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/109 | 2/110 | 1/109
Serious Adverse Events (participants affected / at risk) | 12/109 | 9/110 | 8/109
Other Adverse Events (participants affected / at risk) | 55/109 | 60/110 | 42/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (150 mg Armodafinil) (N=109) | Arm II (250 mg Armodafinil) (N=110) | Arm III (Placebo) (N=109)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (150 mg Armodafinil) (N=109) | Arm II (250 mg Armodafinil) (N=110) | Arm III (Placebo) (N=109)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 4 (4) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (9) | 7 (8) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 3 (3) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (6) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 42 (62) | 46 (67) | 35 (54)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 7 (7) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT01781468/Prot_SAP_001.pdf